CLINICAL TRIAL: NCT04154657
Title: Disclosing Mechanisms of Right Ventricular Adaptation in Patients With Heart Failure With Preserved Ejection Fraction With and Without Pulmonary Hypertension - Insights From Invasive Hemodynamic and Imaging
Brief Title: Mechanisms of Right Ventricular Adaptation in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: INTERACT-HFpEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: University of Giessen (Other)
Responsible Party: Principal Investigator, Birgit Assmus, Director Heart Failure Department, Cardiology, University of Giessen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Interact_HFpEF
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure, Diastolic
Keywords: HFpEF; pulmonary hypertension
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: single cohort observational pathophysiologic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biventricular conductance catheter (Experimental): patients with indication for invasive assessment receive right and left heart catheter and parallel biventricular conductance catheter at rest and stress
  Interventions: Procedure: conductance catheter measurement

INTERVENTIONS:
Procedure: conductance catheter measurement — biventricular parallel conductance catheter measurement at rest and stress conditions, + CMR at rest and stress
  Other Names: pressure volume loop catheter measurement

SUMMARY:
Biventricular PV-loop studies and advanced imaging to assess left-to-right ventricular interaction in HFpEF: In a group of 30 HFpEF patients with clinical indication for LH/RH catheter investigation, we will perform biventricular PV loop assessment in combination with extensive imaging (MRI, echo) for in-depth analysis of left-to-right ventricular interaction in the different HFpEF categories, both under baseline and stress (volume challenge and exercise) conditions.

DETAILED DESCRIPTION:
The right ventricle is the main determinant of prognosis in pulmonary hypertension . The response of the right ventricle to the structural alterations and increasing afterload in the pulmonary circulation is a complex process. The interplay between neuroendocrine and paracrine signalling and increased afterload may lead to myocardial ischemia and inflammation, resulting in loss of myocytes, myocardial fibrosis and RV-arterial uncoupling. Pulmonary hypertension in the setting of heart failure with preserved ejection fraction (HFpEF-PH) is a frequent complication which is associated with impaired prognosis. HFpEF-PH is defined by a high mean pulmonary artery pressure (> 20 mm Hg), high left ventricular end-diastolic pressure (LVEDP > 15 mm Hg) and a normal systolic left ventricular function with impaired diastolic function. However, not all HFpEF patients develop pulmonary vascular remodelling with a high transpulmonary pressure gradient, and increased pulmonary vascular resistance leading to adverse right ventricular remodelling. Ageing, increased left atrial pressure and stiffness, mitral regurgitation, as well as features of metabolic syndrome, including obesity, diabetes and hypertension, are recognized as clinical risk factors for HFpEF-PH. A main and emerging question in that context is the interplay between the right and left ventricle in HFpEF-PH, and whether diastolic left ventricular failure is the driving force of the hemodynamic and right ventricular functional changes. Recent studies have shown that HFpEF-PH patients demonstrate haemodynamic limitations during exercise, including impaired recruitment of LV preload due to excessive right heart congestion and blunted RV systolic reserve compared to HFpEF without PH . However, up to now, no data exist about the mechanism of interplay between RV, LV and pulmonary haemodynamics in HFpEF and HFpEF-PH. Whereas in patients with HFpEF, PV loop analysis has demonstrated that increased end-diastolic pressure at rest is associated with higher end-diastolic stiffness, and a consistently upwards and leftwards shifted pressure volume relationship during exercise and volume challenge, Gortner et al suggest that reduced LV preload (measured by LV transmural pressure gradient) due to excessive RV congestion, is a major driver for reduced cardiac output in HFpEF-PH. However, preliminary own data in 21 patients with HFpEF demonstrate a more complex relationship with approximately one third of patients not showing an increase of (RV and LV ) end-diastolic pressure volume relation during exercise.

Thus, a simultaneous PV loop-catheterization of LV and RV, in addition to right heart catheter, would therefore provide an enormous gain of knowledge about the interaction of RV and LV and would contribute to a better understanding of the pathophysiology of HFpEF-PH and HFpEF.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of HFpEF as follows

* Heart failure NYHA II or NYHA III
* LVEF ≥ 50%
* HFA-PEFF score ≥ 5 OR HFA-PEFF score 2-4 with one of the following criteria:
* baseline PCWP ≥ 15 mm Hg OR PCWP increase ≥ 10 mm Hg with exercise (~20 Watt)
* stable medical therapy for last 4 weeks

Exclusion criteria:

* Significant coronary stenosis > 50% or valvular heart disease requiring intervention
* coronary or cardiac valvular intervention < 3 months
* uncontrolled rate of atrial fibrillation
* Severe chronic kidney disease (MDRD eGFR < 30 ml/min)
* Life expectancy < 12 months
* Contraindication to MRI or other planned investigations

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
delta Eed | immediate after procedure
  RV stiffness measured by conductance catheter is reduced alreday in early HFpEF stages
delta RV volume | immediate after procedure
  homeometric followed by teterometric adaptation with consecutive dilation of the RV occurs with disease progression from HFpEF-Non-PH ti ICC-PH_HFpEF to cpc-PH-HFpEFprogressive H, impacting position and motion of the septum with stress

SECONDARY OUTCOMES:
correlation of delta RV longitudinal strain with Eed | immediate after procedure
  RV longitudinal strain (related to RV EDV) is the best predictor of RV diastolic stiffness (Eed) in HFpEF-PH (correlation analysis)
delta transmural septal pressure | immediate after procedure
  acute change of the transmural pressure gradients from rest to stress conditions, adversly impacts LV filling

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Goethe University Hospital, Frankfurt am Main, Hesse
  - University Hospital Justus-Liebig University, Giessen

IPD SHARING:
Plan to Share IPD: No